CLINICAL TRIAL: NCT01081626
Title: A Phase IV, Open-label, Post Marketing, Prospective, Randomized, Controlled, Multicentre, Multinational Study to Investigate Tailoring of Recombinant FSH Use in Ovulation Stimulation Treatment in Chronic Anovulatory Subjects (WHO Group II)
Brief Title: Recombinant Follicle Stimulating Hormone (FSH) (Gonal-f®): Use in Ovulation Induction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono Middle East FZ-LLC, United Arab Emirates, an affiliate of Merck KGaA, Darmstadt, Germany (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMR 700623-501
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Results first posted 2012-11-07 (Estimated); Last update posted 2014-02-13 (Estimated); Status verified 2014-01

CONDITIONS: Ovulation Induction
Keywords: Infertility; Ovulation induction; Gonal-f; Follitropin alpha; Polycystic ovarian syndrome; Anovulatory infertility
MeSH Terms: conditions — Infertility; Polycystic Ovary Syndrome | interventions — Glycoprotein Hormones, alpha Subunit; follitropin alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group I: Chronic Low dose Protocol (Experimental): Gonal-f will be injected on the second or third day of a spontaneous or progestogen-induced menstrual cycle (Day 0), with a daily dose of 75 International Units (IU) for 7 days. Ovarian response will be assessed on Day 7 of stimulation by ultrasound scan. If no follicle has reached at least 10 to 12 millimeter (mm) diameter, stimulation will be continued with the same dose for further 7 days. On Day 14 of stimulation, if no ovarian response is seen, the dose will be increased by 37.5 IU (total 112.5 IU) and administered for the next 7 days. Subsequent increments of 37.5 IU, at intervals of 7 days up to Day 35 of stimulation would be made, depending on ovarian response.
  Interventions: Drug: Recombinant FSH (follitropin alpha)
- Group II: Low dose Protocol (Experimental): Gonal-f will be administered on the second or third day of a spontaneous or progestogen-induced menstrual cycle (Day 0), with a daily dose of 75 IU for 7 days. Ovarian response will be assessed on Day 7 of stimulation by ultrasound scan. If no follicle has reached at least 10 to 12 mm diameter, the dose will be increased by 37.5 IU (total 112.5 IU) and administered for the next 7 days. Subsequent increments of 37.5 IU, at intervals of 7 days up to Day 35 of stimulation will be made, depending on ovarian response.
  Interventions: Drug: Recombinant FSH (follitropin alpha)

INTERVENTIONS:
Drug: Recombinant FSH (follitropin alpha) — A starting dose of 75 IU and a first adjustment on Day 14 or Day 7 of stimulation in Group I and II respectively, if no ovarian response is observed.
  Other Names: Gonal-f®; Follitropin alpha

SUMMARY:
This is an open-label, prospective, randomized, controlled, multicentric, multinational, phase IV study to evaluate the use of Gonal-f in inducing ovulation in female subjects with chronic anovulation. It has been observed that conventional high dose set up regimen of gonadotropin and human chorionic gonadotropin (hCG) is effective in anovulatory subjects in terms of overall pregnancy rates. However, development of multiple follicles leading to multiple pregnancy and/or ovarian hyperstimulation syndrome (OHSS) is the major complications associated with this high dose set up. Chronic low-dose (CLD) protocols of follicle stimulating hormone (FSH), aimed at finding the threshold amount of FSH necessary to promote monofolliculogenesis, have been found to be successful in reducing the rate of OHSS almost to nil and the rate of multiple pregnancies to a minimum. This post-marketing study will investigate tailoring of recombinant follicle stimulating hormone (r-FSH) in a large population (N=310) of subjects from a region (North Africa/Middle East) that has not been included in previous studies of ovulation induction in subjects with chronic anovulation. The study aims to increase current knowledge of the efficacy and safety of Gonal-f, and provide fertility physicians with experience in Gonal-f treatment in anovulatory infertility, thereby contributing to the development of FSH dosing guidelines for ovulation induction by defining the optimal CLD and Low dose (LD) regimens.

DETAILED DESCRIPTION:
Gonal-f is a recombinant form of human FSH (r-hFSH), an endogenous gonadotropin which is being produced in genetically engineered chinese hamster ovary cells and is indicated for induction of ovulation and pregnancy in anovulatory infertile women in whom the cause of infertility is functional and not due to primary ovarian failure. It is also indicated for the development of multiple follicles in ovulatory women participating in an assisted reproductive technology (ART) programme, such as in in vitro fertilization (IVF). The primary cause of infertility in women is an abnormality of ovulation. Most of these anovulatory subjects fall into the World Health Organization (WHO) Group II category, characterized by asynchronous gonadotropin and oestrogen production and normal levels of prolactin (PRL). These subjects present with a variety of menstrual disorders, most commonly polycystic ovarian syndrome (PCOS).

Gonal-f is administered as a course of daily injections, subcutaneously into the anterior abdominal wall. A commonly used regimen commences at 75-150 IU FSH daily and is increased preferably by 37.5 IU, or 75 IU at 7 or preferably 14 day intervals if necessary, to obtain an adequate but not excessive response. A single injection of 5,000 IU urinary hCG (u-hCG) (or 250 microgram [mcg] r-hCG) should be administered after the last dose of Gonal-f and when the leading follicle has reached 17 mm in diameter. The subject is later recommended to have coitus on the day of, and the day following, hCG administration. The efficacy of Gonal-f in the treatment of WHO Group II anovulatory infertile women has been confirmed by 2 randomized, open-label, multicentric, phase III non-inferiority studies that compared Gonal-f with Metrodin® (urinary FSH) for ovulation induction. The possible serious adverse events (SAEs) associated with Gonal-f include OHSS and its possible complications, multiple pregnancies, pregnancy wastage, ectopic pregnancies and the possible risk of ovarian cancer and reproductive system neoplasms (e.g. endometrial, breast carcinoma).

OBJECTIVES

Primary objective:

* To investigate tailoring of recombinant FSH treatment in subjects with chronic anovulation

Secondary objectives:

* To evaluate commonly used ovulation induction regimens and treatments
* To establish local experience with the Gonal-f pen and investigate ease of use

The study will enroll 310 eligible subjects, randomized in a 1:1 ratio to either Group I or II at the baseline visit prior to the first dose of FSH (pre-stimulation). Each subject will be refrained from the use of gonadotropins or any other ovulation stimulation therapy during the period from screening to the start of stimulation treatment. During the stimulation period, Gonal-f will be administered as a course of once daily (OD) injections, s.c. into the anterior abdominal wall through Gonal-f pen, according to either one of the following 2 step-up, low-dose regimens:

Group I: CLD regimen which recommends a starting dose of 75 IU and a first adjustment on Day 14 of stimulation, if no ovarian response is observed.

Group II: LD regimen which recommends a starting dose of 75 IU and a first adjustment on Day 7 of stimulation, if no ovarian response is observed.

For both groups, when at least 1 follicle reaches 10 to 12 mm in diameter, the Gonal-f administration will be maintained at that dose until the leading follicle reaches 17 mm or more in diameter and no more than 2 follicles have reached 14 mm in diameter. A single injection of hCG (5,000 IU u-hCG or 250 mcg r-hCG) will be administered intramuscularly or subcutaneously after the last Gonal-f injection, to trigger ovulation. Subjects will also be advised to have coitus on the day of, and the day following hCG administration. The total length of the stimulation treatment will not exceed 35 days unless an ultrasound assessment suggests imminent follicular growth and maturation and each subject will undergo one cycle of stimulation treatment only. Subjects will also be followed for a post stimulation period of up to 20 days after the triggering of ovulation by hCG injection, or cancellation of the cycle.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal female subjects, aged between 18 and 37 years inclusive
* Subjects willing to conceive
* Subjects who are infertile due to chronic anovulation demonstrated by a cycle duration of > 35 days, or regular cycles with progesterone (P4) levels < 1 nanomole/milliliter (nmol/mL) during luteal phase (Day 25)
* Subjects who have experienced spontaneous menses, menses induced by clomiphene citrate therapy, or a positive progestin-induced withdrawal within the previous year
* Subjects with FSH and PRL serum values within the normal range in the early follicular phase
* Subjects with total antral follicle count (AFC) > 10 (of follicle size ≥ 2 mm and < 11 mm) in both ovaries
* Subjects with at least 1 patent tube, as documented by recent (within 2 years before treatment assignment) hysterosalpingography (HSG)
* Subjects with normal uterine cavity, as documented by recent (within 2 years before treatment assignment) hysteroscopy, HSG or ultrasound scan
* Subjects with body mass index (BMI) >20 and ≤32 kilogram square per meter (kg/m^2)
* Subjects with negative cervical Papanicolaou (PAP) test within the 6 months prior to screening
* Male partners of female subjects with sperm compatible with non assisted fertilization
* Subjects who are willing and able to participate in the study and have provided written, informed consent

Exclusion Criteria:

* Subjects with history of hypersensitivity to the active substance follitropin alpha, FSH, or to any of the excipients of Gonal-f
* Subjects with ovarian enlargement or ovarian cyst unrelated to PCOS, and of unknown origin on ultrasound
* Subjects with evidence of diminished ovarian reserve (cycle length < 26 days; FSH above the upper limit of local serum FSH values, total AFC in both ovaries < 10)
* Subjects with myomatous uterus, which in the opinion of the investigator could impair pregnancy evolution
* Subjects who have undergone 3 or more previous miscarriages
* Subjects with any previous extrauterine pregnancy
* Pregnant or lactating female subjects
* Subjects with abnormal gynecological bleeding of unknown etiology
* Subjects with previous history of severe OHSS
* Subjects who have undergone operative pelvic surgery which could induce mechanical infertility (e.g tubes blockage) or pelvic inflammatory disease (PID) before treatment assignment excluding curettage and hysteroscopy
* Subjects with tumors of the hypothalamus and pituitary gland
* Subjects with ovarian, uterine or mammary carcinoma
* Subjects treated with clomiphene citrate or gonadotropins within 1 month of the screening evaluation
* Subjects with any medical condition which, in the opinion of the investigator, would prevent an effective response, such as primary ovarian failure, or malformations of the reproductive organs incompatible with pregnancy
* Subjects with any medical condition which, in the opinion of the investigator, may interfere with the absorption, distribution, metabolism or excretion of the drug
* Subjects with any clinically significant systemic disease (e.g. insulin-dependent diabetes) or any contraindication to being pregnant and/or carrying a pregnancy to term; also including subjects with non insulin dependent diabetes mellitus (NIDDM)
* An active substance abuser
* Subjects with known infection with Human Immunodeficiency Virus (HIV), Hepatitis B or C virus in the trial subject or her male partner
* Subjects who have simultaneously participated in another clinical trial

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 310 (Actual)
Dates: Start 2009-03; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Esmat, MD, Study Director — Merck Serono Middle East FZ-LLC, United Arab Emirates, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (3):
- New Mowasat Hospital, As Sālimīyah, P.O.Box 6661, Kuwait
- Mount Lebanon Hospital, Hazmiyeh, P.O.Box 470, Lebanon
- King Abdel Aziz University Hospital, Jeddah, P.O.Box 80215, Saudi Arabia

REFERENCES:
- [Derived] Serour GI, Aboulghar M, Al Bahar A, Hugues JN, Esmat K. Phase IV, open-label, randomized study of low-dose recombinant human follicle-stimulating hormone protocols for ovulation induction. Reprod Biol Endocrinol. 2014 Jun 18;12:52. doi: 10.1186/1477-7827-12-52. PMID 24942155

RESULTS

PARTICIPANT FLOW:
Groups:
- Chronic Low Dose (CLD) Protocol: Gonal-f® (follitropin alpha) injection 75 International Units (IU) subcutaneously administered for 7 days. Dose increased by 37.5 IU on Day 14 of stimulation period, at intervals of 7 days up to Day 35 of stimulation period or until ovarian response observed.
- Low Dose (LD) Protocol: Gonal-f® (follitropin alpha) injection 75 IU subcutaneously administered for 7 days. Dose increased by 37.5 IU on Day 7 of stimulation period, at intervals of 7 days up to Day 35 of stimulation period or until ovarian response observed.
Period: Overall Study
Arm/Group | Chronic Low Dose (CLD) Protocol | Low Dose (LD) Protocol
Started | 155 | 155
Assessed for Efficacy | 122 | 125
Completed | 95 | 94
Not Completed | 60 | 61
Not completed — Dosing error | 1 | 1
Not completed — Missing Estradiol | 25 | 28
Not completed — Low antral follicle count | 1 | 0
Not completed — Overstimulation | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Other | 33 | 30

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chronic Low Dose (CLD) Protocol | Low Dose (LD) Protocol | Total
Number analyzed (Participants) | 122 | 125 | 247
Age, Continuous [Mean (Standard Deviation); unit: years] — Data for baseline measure (age) was available for 122 and 125 participants in CLD protocol and LD protocol arm, respectively, who were treated and had at least 1 efficacy evaluation.
  years | 27.51 (4.42) | 27.88 (4.33) | 27.70 (4.37)
Sex: Female, Male [Count of Participants; unit: Participants] — Data for baseline measure (gender) was available for 122 and 125 participants in CLD protocol and LD protocol arm, respectively, who were treated and had at least 1 efficacy evaluation.
  Participants
    Female | 122 | 125 | 247
    Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Mono-follicular Development
Description: Mono-follicular development was defined as the development of only 1 follicle of greater than or equal to (>=) 17 millimeter (mm) diameter and no more than 2 other follicles larger than 14 mm in diameter at or before Days 35-42 of stimulation period assessed by means of a transvaginal ultrasound scan.
Time Frame: Day 0 (first dose) up to Days 35-42 post human chorionic gonadotropin [hCG] administration (end of stimulation cycle {less than or equal to [<=] 35 days})
Population: The Intention-To-Treat (ITT) population included all the participants who received at least 1 dose of study medication, had 1 efficacy assessment and did not have any protocol criteria violations or did not receive a wrong treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Chronic Low Dose (CLD) Protocol | Low Dose (LD) Protocol
Number analyzed (Participants) | 122 | 125
percentage of participants | 56.55 | 55.20
Statistical Analysis 1: Comparison: Chronic Low Dose (CLD) Protocol vs Low Dose (LD) Protocol; Test type: Superiority or Other; p = 0.9560, Chi-squared, Corrected; Mean Difference (Final Values) = 0.0135, 95% CI 2-sided [-0.1325 to 0.1637]

2. Secondary Outcome: Number of Participants With Multi-follicular Development
Description: Multi-follicular development was defined as the development of more than 3 follicles >= 15 mm in diameter at or before Days 35-42 of stimulation period assessed by means of a transvaginal ultrasound scan.
Time Frame: Day 0 (first dose) up to Days 35-42 post hCG administration (end of stimulation cycle {less than or equal to [<=] 35 days})
Population: The ITT population included all the participants who received at least 1 dose of study medication, had 1 efficacy assessment and did not have any protocol criteria violations or did not receive a wrong treatment.
Measure: Number; unit: participants
Arm/Group | Chronic Low Dose (CLD) Protocol | Low Dose (LD) Protocol
Number analyzed (Participants) | 122 | 125
participants | 17 | 15
Statistical Analysis 1: Comparison: Chronic Low Dose (CLD) Protocol vs Low Dose (LD) Protocol; Test type: Superiority or Other; p = 0.7924, Chi-squared; Risk Ratio (RR) = 1.088, 95% CI 2-sided [0.7642 to 1.5490]

3. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: AE: any new untoward medical occurrence/worsening of pre-existing medical condition, whether or not related to study drug.
Time Frame: as for outcome 2
Population: The safety population included all the participants who received at least 1 dose of study medication and had 1 follow-up visit.
Measure: Number; unit: participants
Arm/Group | Chronic Low Dose (CLD) Protocol | Low Dose (LD) Protocol
Number analyzed (Participants) | 155 | 155
participants | 30 | 31

4. Secondary Outcome: Number of Participants With Multiple Pregnancies
Description: Multiple pregnancy is a pregnancy where more than one fetus develops simultaneously in the womb. There are two types of twinning-identical and fraternal. Identical twins represent the splitting of a single fertilized zygote (union of two gametes or male/female sex cells that produce a developing fetus) into two separate individuals.
Time Frame: as for outcome 2
Population: The ITT population included all the participants who received at least 1 dose of study medication, had 1 efficacy assessment and did not have any protocol criteria violations or did not receive a wrong treatment. Number of participants analyzed (N) included participants who were evaluated for this particular measure.
Measure: Number; unit: participants
Arm/Group | Chronic Low Dose (CLD) Protocol | Low Dose (LD) Protocol
Number analyzed (Participants) | 94 | 91
participants | 3 | 1

5. Secondary Outcome: Number of Participants With Injection Tolerability
Description: Participants who did not show any injection site reactions such as pain, redness, bruises, swelling and irritation were considered to have injection tolerability.
Time Frame: as for outcome 2
Population: The safety population included all the participants who received at least 1 dose of study medication and had 1 follow-up visit. Number of participants analyzed (N) included participants who were evaluated for this particular measure.
Measure: Number; unit: participants
Arm/Group | Chronic Low Dose (CLD) Protocol | Low Dose (LD) Protocol
Number analyzed (Participants) | 73 | 77
participants | 54 | 54

6. Secondary Outcome: Number of Participants Who Received Human Chorionic Gonadotropin (hCG)
Time Frame: End of stimulation cycle (less than or equal to [<=] 35 days)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Chronic Low Dose (CLD) Protocol | Low Dose (LD) Protocol
Number analyzed (Participants) | 122 | 125
participants | 94 | 91
Statistical Analysis 1: Comparison: Chronic Low Dose (CLD) Protocol vs Low Dose (LD) Protocol; Test type: Superiority or Other; p = 0.5331, Chi-squared

7. Secondary Outcome: Number of Participants With Cancelled Cycles
Description: Participants with cancelled cycles were those who did not achieve adequate follicular formation (at least 17 mm) for hCG administration.
Time Frame: End of stimulation cycle (less than or equal to [<=] 35 days)
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Chronic Low Dose (CLD) Protocol | Low Dose (LD) Protocol
Number analyzed (Participants) | 122 | 125
participants | 19 | 19
Statistical Analysis 1: Comparison: Chronic Low Dose (CLD) Protocol vs Low Dose (LD) Protocol; Test type: Superiority or Other; p = 0.9351, Chi-squared; Risk Ratio (RR) = 1.015, 95% CI 2-sided [0.7175 to 1.4350]

8. Secondary Outcome: Number of Participants With Clinical Pregnancies
Description: Clinical pregnancy was defined as pregnancy diagnosed by ultrasonographic visualization of one or more gestational sacs or definitive clinical signs of pregnancy. It includes ectopic pregnancy.
Time Frame: as for outcome 2
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Chronic Low Dose (CLD) Protocol | Low Dose (LD) Protocol
Number analyzed (Participants) | 94 | 91
participants | 19 | 18

9. Secondary Outcome: Duration of Follicle Stimulating Hormone (FSH)
Time Frame: End of stimulation cycle (less than or equal to [<=] 35 days)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Chronic Low Dose (CLD) Protocol | Low Dose (LD) Protocol
Number analyzed (Participants) | 94 | 91
Days | 13.68 (6.33) | 12.85 (5.58)

10. Secondary Outcome: Total Follicle Stimulating Hormone (FSH) Dose
Time Frame: End of stimulation cycle (less than or equal to [<=] 35 days
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: IU
Arm/Group | Chronic Low Dose (CLD) Protocol | Low Dose (LD) Protocol
Number analyzed (Participants) | 94 | 91
IU | 1119.41 (690.04) | 1155.47 (730.45)

11. Secondary Outcome: Number of Participants Who Answered Ease of Use of Gonal-f® Pen Questionnaire
Description: Ease of use of Gonal-f® pen was assessed through a questionnaire consisting of 23 questions and the number of participants who responded to the questionnaire was recorded.
Time Frame: On hCG administration day (end of stimulation cycle {less than or equal to [<=] 35 days})
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Chronic Low Dose (CLD) Protocol | Low Dose (LD) Protocol
Number analyzed (Participants) | 122 | 125
participants | 58 | 75

ADVERSE EVENTS:
Time Frame: AEs were collected on an ongoing basis from day of written informed consent. All new AEs were recorded until the post-treatment safety, on day 35-42 post-hCG administration.
Description: Pre-Treatment:Medical conditions present at the initial study visit that did not worsen in severity or frequency during the study;Treatment-Emergent: If the onset date of the AE was on or after the first dose date of the study medication; Post-Treatment: If the onset date of the AE was post-hCG Days 35- 42 for participants who completed the study.
Arm/Group | Chronic Low Dose (CLD) Protocol | Low Dose (LD) Protocol
Serious Adverse Events (participants affected / at risk) | 0/155 | 1/155
Other Adverse Events (participants affected / at risk) | 30/155 | 30/155
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chronic Low Dose (CLD) Protocol (N=155) | Low Dose (LD) Protocol (N=155)
Ectopic pregnancy (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chronic Low Dose (CLD) Protocol (N=155) | Low Dose (LD) Protocol (N=155)
Dizziness (Cardiac disorders) | 1 | 5
Burning pain of the stomach (Gastrointestinal disorders) | 0 | 1
Abdominal colic pain (Gastrointestinal disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 12 | 7
Gums swelling (Gastrointestinal disorders) | 0 | 1
Heart burn (Gastrointestinal disorders) | 0 | 1
In abdomen (Gastrointestinal disorders) | 0 | 1
Lower abdominal pain (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 5 | 5
Pain in stomach (Gastrointestinal disorders) | 0 | 4
Vomiting (Gastrointestinal disorders) | 0 | 1
Abdominal bloating (Gastrointestinal disorders) | 1 | 0
Burning (General disorders) | 1 | 0
Fever (General disorders) | 2 | 0
Generalized fatigability (General disorders) | 1 | 0
Pain (General disorders) | 2 | 0
Spasm and pain (General disorders) | 1 | 0
Chest pain (General disorders) | 0 | 3
Fatigue (General disorders) | 0 | 1
Hot flash (General disorders) | 0 | 1
Allergic rhinitis (Immune system disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3
Joint pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in the foot (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in the right loin (Musculoskeletal and connective tissue disorders) | 1 | 0
Legs pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Lower back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Weakness Generalized (Musculoskeletal and connective tissue disorders) | 0 | 1
Body pain (General disorders) | 0 | 1
Headache (Nervous system disorders) | 10 | 14
Drowsiness (Psychiatric disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 1 | 1
Nervousness (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Lethargy (Psychiatric disorders) | 0 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 1
Ectopic pregnancy (Reproductive system and breast disorders) | 0 | 1
Ovarian Hyper Stimulation Syndrome (Reproductive system and breast disorders) | 1 | 0
Blood (General disorders) | 0 | 1
Car accident (spotting) (General disorders) | 1 | 0
Cold (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Itching in upper and lower limb and abdomen (Skin and subcutaneous tissue disorders) | 1 | 0
Insect bite (Skin and subcutaneous tissue disorders) | 0 | 1
Itching (Skin and subcutaneous tissue disorders) | 0 | 1
Itching and burning (Skin and subcutaneous tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other